CLINICAL TRIAL: NCT04523155
Title: Effect of Medically-tailored Meal Delivery Service on Changes in Hemoglobin A1c (HbA1c) in Patients With Diabetes: A Randomized, Crossover Clinical Trial
Brief Title: Effect of Medically-tailored Meal Delivery Service on Changes in Hemoglobin A1c (HbA1c) in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Farford, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-004608
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants randomized to sequence AB will receive 3 months of meals, followed by a 3 month washout period and a 3 month intervention period with no meals.
  Interventions: Dietary Supplement: Medically tailored meals
- Treatment Sequence BA (Experimental): Participants randomized to sequence BA will receive 3 months of no meals followed by a 3 month washout period and a 3 month intervention period with meals.
  Interventions: Dietary Supplement: Medically tailored meals

INTERVENTIONS:
Dietary Supplement: Medically tailored meals — 10 meals per week for 3 months

SUMMARY:
The purpose of this study is to evaluate the effect of medically-tailored meal delivery (10 meals per week for 3 months) on glycemic control in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women with non-insulin dependent diabetes.
* Ages 25 to 75 years.
* Fasting blood sugar of greater than 140 mg/dl, on no oral hypoglycemic agents and a hemoglobin A1C less than 13%.
* Stabilized patients on oral hypoglycemic agents for one month or longer prior to starting the study and a hemoglobin A1C between 7.5% - 13%.

Exclusion Criteria:

* Insulin use.
* Substance abuse.
* Any documented medical problem that would inhibit full participation in the study.
* BMI less than 25 or great than 40.
* Vegans or Vegetarians
* Individuals with food allergies.
* Individuals currently on a commercial weight loss or diet program.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Change in Glucose Metabolism | Baseline, 3 monts
  Measured by HbA1c levels in standard chemistry in blood

SECONDARY OUTCOMES:
Change in Weight | Baseline, 3 months
  Measured in killograms
Change in Blood Pressure | Baseline, 3 months
  Measured in units of millimeters of mercury (mmHg)
Change in High Density lipoprotein (HDL) | Baseline, 3 months
  HDL cholesterol levels measured by standard chemistry in blood reported in units of milligrams per deciliter (mg/dL)
Change in Low Density Lipoprotein (LDL) | Baseline, 3 months
  LDL cholesterol levels measured by standard chemistry in blood reported in units of milligrams per deciliter (mg/dL)
Change in Triglycerides | Baseline, 3 months
  Triglyceride levels measured by standard chemistry in blood reported in units of milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Farford, DO, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials